CLINICAL TRIAL: NCT00471913
Title: Functional Outcome and MR Imaging of Abductor Damage Following Antegrade Femoral Nailing With Different Entry Points: A Prospective Randomized Trial
Brief Title: Functional Outcome and MRI of Muscle Damage Following Nailing Procedure in Femur (Thigh) Fractures Using Different Entry Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Pierre Guy, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H06-03242
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Femoral Shaft Fracture
Keywords: Femur; Fracture; Antegrade; Nailing; Shaft; Abductor
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Femoral Nailing with Different Entry Points — See Detailed Description.

SUMMARY:
Study focus is femoral shaft (thigh bone) fractures (break) that require surgical treatment under anaesthetic to stabilize the femur fracture. This is usually done by placing a metal nail and screws inside the femur (thigh) bone.

This study has been designed to allow us to learn more about the effect of using a different starting point to insert the nail into the body in order to access the fracture and fix it. This question is important because to date, all entry points currently used do result in some muscle damage. In order to minimize this damage a lateral (side) entry nail has been developed and is currently in use at many centres. This nail is new but, the lateral entry technique for these types of fractures has been used extensively in the past, and this nail has been developed in order to better accommodate the technique.

It is believed that entering laterally instead of going deeper into the tissue to access the bone to fix it is going to result in less muscle damage which in turn will improve functional outcome.

DETAILED DESCRIPTION:
Background:

This study has been designed to prospectively evaluate functional outcome and MR imaging of abductor damage following antegrade femoral nailing with different entry points

Recent developments in IM nailing of the femur have favoured the use of the greater trochanter as an entry site as opposed to using the "classical" piriformis fossa. With either technique, a persistent problem appears however to be the damage caused to muscle tissue during preparation of the femur and insertion of the nail. The recent development of femoral nails with an entry point lateral to both these sites offers the potential advantage of avoiding abductor muscle damage.

In several cadaver studies, authors state that a trochanteric entry point causes more damage than a piriformis entry, and that an even more lateral entry point causes even less damage to the abductor muscles compared to the classical piriformis fossa entry site. There is however, no prospective clinical study has specifically evaluated the condition of the abductor tendon and the amount of muscle damage after antegrade nailing in the treatment of femoral shaft fractures. The few clinical studies that have attempted to examine the functional outcome in patients undergoing IM nailing of femoral fractures have used general measurement tools (general functional clinical assessment, gross evaluation of gait) which do not reflect the state of the art at this time and which do not specifically assess gluteal muscle condition. To date, no published study has evaluated the integrity of the gluteus tendon, the damage to the surrounding tissues, and the functional outcome using validated scores. Moreover, no study has compared the "traditional" entry points to a lateral entry nail with this level of precision.

The standard of care for the treatment of femoral shaft fractures is the insertion of an intramedullary nail through the piriformis fossa. Following insertion of femoral IM nails, a number of studies have demonstrated excellent clinical and radiographic results with relatively few complications such as nonunion, malunion, or infection. Intraoperative difficulties with respect to rapid identification of the appropriate starting point have prompted the development of nails that use the greater trochanter as an entry site as opposed to using the "classical" piriformis fossa.

As stated earlier, with either technique, a persistent problem appears however to be the damage caused to muscle tissue during preparation of the femur and insertion of the nail. The recent development of femoral nails with an entry point lateral to both these sites offers the theoretical advantage of avoiding abductor muscle damage. There is so far a lack of prospective randomized trials which demonstrate radiological and clinical parameters of the different entry points.

Objective To determine the abductor tendon and muscle damage with MR-imaging according to the entry point of the femoral nail. Additionally, objective hip muscle function, general health status and functional outcome will be assessed using validated instruments.

We aim to correlate muscle damage due to the different entry points and correlate with the functional outcome. Further, to quantify the differences (advantages) of different IM nailing techniques of the femur, with respect to effect on the abductor musculature, muscle testing and gait, and patient-based functional outcome, to guide surgeons' decisions and future research.

Recent Related Work In a recently published report by Ricci et al. the use of the trochanteric entry point was associated with a low complication rate and good clinical results including the assessment of a gait video. In this admittedly small prospective study the superiority of either the trochanteric or the piriformis fossa entry point nail could not be established. Although gait was evaluated video (in 30% of the study population), this was limited to a subjective assessment of the presence of a Trendelenberg gait (absent, slight or present). There was no statement about the muscle status, and functional outcome assessment was limited to a Harris Hip Score.

Abductor tendon condition and muscle damage has previously been assessed with MR-imaging by the group of Pfirrmann et al. in patients with total hip arthroplasty through a transgluteal approach. This study showed a high correlation between damage and clinical outcome.

The co-applicant's research group has previously carried out many clinical studies including its part in a multi-centre randomized trial in femur fractures. It also specifically has carried out a functional assessment of patients following femur fractures which included: objective muscle testing of isokinetic force using a KinCom® dynamometer, formal gait lab analysis using an eight camera real-time motion capture system in conjunction with a force-plate walking platform, and as part of the same study, the administration of validated self-assessment outcome questionnaires.

So far no prospective randomized trial has investigated, as we have planned to do, the radiological (MR), functional, and clinical outcome after insertion of a femoral nail through two different entry points.

Method Patients will be assigned randomly (via computer generated randomization) to one of two groups. The two groups will undergo standard treatment of IM nailing for the femoral shaft fracture differing only in entry point of the nail: piriformis fossa entry point versus lateral entry point.

Design Patients between 19 and 60 years of age presenting with an isolated femoral shaft fracture that requires IM nailing will be asked to participate in this study. Informed consent for participation in the study will be obtained by either a member of the health care team or by a research nurse.

Consenting patients who meet the inclusion criteria will be randomized to either piriformis fossa or lateral entry femoral nailing. Preoperative, Intraoperative, and follow-up data will be obtained. Data will detail clinical assessment, MRI results, objective muscle testing, and gait analysis.

Power analysis In a published report from Pfirrmann et al. distinct conclusions could be made in a collective of 54 patients. We plan to recruit 60 patients (30 per group) with a projected drop-out rate of 10%. As this is a pilot study, without previous reference, a similarity in expected findings and required sample size must be inferred. Cases will be randomized using a web-based allocation tool.

Outcome Variables:

Variables for collection and analysis are:

1. Preoperative:

   i) Demographics ii) ISS (Injury Severity Score) iii) AO Fracture Classification
2. Intraoperative:

   i) Elapsed time from injury to operative treatment ii) Fluoroscopy time iii) Incision length iv) Blood loss
3. Postoperative:

   i) VAS pain scores ii) Morphine requirements q 24hrs iii) Change in hemoglobin q 24hrs iv) Hospital Length of Stay v) Clinical and Radiological follow-up at 3, 6, 9, and 12 months vi) MRI at 12 months vii) Self-administered validated outcome tools at 6 and 12 months (SF-36, SMFA, Harris Hip Score, Merle d'Aubigne score) although last two are not validated they would allow for comparison with widely published scores in established literature

   Study Specific Measures:

   Postoperative follow-up:

   All patients will be reviewed clinically in the fracture clinic at two, six, twelve weeks, and six and twelve months postoperatively. Study data will be acquired at the six and 12 month appointments.

   Clinical assessment:

   Bilateral measurements will be recorded so that the results from the unaffected limb are used as a control for the injured limb. Both the raw data and the side to side differences will be used in the analysis. Physical examination to document any limb length discrepancy, Trendelenberg sign, rotational malalignment, and the ranges of motion of the hip and knee.

   Questionnaires:

   A study specific questionnaire will be administered to determine the extent and location of any persistent pain in the affected limb, ability to return to their usual occupation and recreational activities.

   Functional outcome scores (SF-36, SMFA, Harris Hip Score, Merle d'Aubigne score) will be collected at 6 and 12 months. All of these outcomes tools are widely referenced in the literature and can be used for comparison purposes.

   MR Imaging:

   An MRI will be administered at 12 months and will include evaluation of abductor tendon defects, diameter, signal intensity, ossification, and bursal fluid collections. The abductor muscles will be evaluated by MRI for fatty atrophy.

   Muscle strength testing and gait analysis:

   Muscle strength testing will take place at 12 months and will utilize the KinCom Dynamometer (a widely used, standard research protocol and specifically-designed instrument for use in muscle strength testing) to evaluate muscle strength: Peak isokinetic force measurement: maximum strength (nm/kg), and work (J/min) of hip abductors, hip extensors, and knee extensors.

   Gait analysis will take place at 12 months and will employ a standard eight camera real-time motion capture system in conjunction with a force-plate walking platform to collect and evaluate pelvic obliquity, hip abductor movement, single leg support time, and step length.

   Data Analysis:

   The side-to-side differences will be summarized and compared across treatment groups. Additionally, aggregated raw data by treatment group will be summarized and compared, using t-test for the comparison of continuous variables' means, and Chi-square for categorical data.

ELIGIBILITY:
Inclusion Criteria:

* 19 to 60 years of age
* Isolated closed femoral shaft fracture
* Ability to take part in follow-up and functional testing

Exclusion Criteria:

* Patients under 19 and over 60 years of age
* Non - traumatic/pathological fractures
* Ipsilateral acetabulum/pelvis fracture
* Open femoral shaft fracture
* Previous lower extremity surgery
* Pre-existing disability
* Presents for revision surgery
* Mentally incompetent to consent

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
12 month functional outcome and determination of muscle and tendon damage with MR Imaging | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Guy, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada